CLINICAL TRIAL: NCT05690087
Title: Effect of Systemic Lidocaine Infusion on Optic Nerve Sheath Diameter in Patients Undergoing Laparoscopic Hysterectomy in Trendelenburg Position
Brief Title: Lidocaine Infusion on Optic Nerve Sheath Diameter in Laparoscopic Hysterectomy in Trendelenburg Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Osama Rehab, Lecturer of Anesthesiology, Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36204/12/22
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-03

CONDITIONS: Lidocaine; Optic Nerve Sheath Diameter; Laparoscopic Hysterectomy; Trendelenburg
MeSH Terms: interventions — Lidocaine; Sodium Chloride; Solutions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine group (Experimental): Intravenous lidocaine 2% bolus of 1.5 mg/kg over 5 min before induction of anesthesia followed by lidocaine infusion at 1.5 mg/kg/h intraoperatively until desufflation.
  Interventions: Drug: Lidocaine
- Control group (Placebo Comparator): Intravenous sodium chloride 0.9% solution volume matched in bolus and infusion.
  Interventions: Drug: sodium chloride 0.9% solution

INTERVENTIONS:
Drug: Lidocaine — intravenous lidocaine 2% bolus of 1.5 mg/kg over 5 min before induction of anesthesia followed by lidocaine infusion at 1.5 mg/kg/h intraoperatively until desufflation
  Arms: Lidocaine group
Drug: sodium chloride 0.9% solution — intravenous sodium chloride 0.9% solution volume matched bolus and infusion.
  Arms: Control group

SUMMARY:
We hypothesize that intravenous lidocaine infusion may have beneficial effect to patients undergoing laparoscopic surgeries in Trendelenburg position by preventing ICP elevation.

DETAILED DESCRIPTION:
Lidocaine use, both intravenous (IV) and laryngotracheal (LT), has been reported to blunt the ICP elevations during intubation. Also, Lidocaine injected IV has been shown in models to induce cerebral vasoconstriction leading to a decrease in cerebral blood volume and thus ICP. Furthermore, IV lidocaine leads to sodium channel inhibition and thus a reduction in cerebral activity and metabolic demands, as well as excitotoxicity, leading to a potential ICP reduction effect.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 35 to 65 years
* American society of anesthesiology (ASA) physical status I - II
* Body mass index (BMI) between 18.5 to 28.0 kg/m2
* Scheduled for total laparoscopic hysterectomy taking approximately 2 h with a 30° Trendelenburg position for management of uterine fibroids or refractory dysfunctional uterine bleeding.

Exclusion Criteria:

1. Patients with eye diseases, central nervous system diseases, cardiovascular diseases, cerebrovascular diseases or diabetes.
2. If these events occurred intraoperative:

   * Ultrasound scans or measurements failed to clearly show the structure of Optic Nerve Sheath Diameter (ONSD).
   * Surgical time less than 1 h.
   * Interruption of carbon dioxide (CO2) pneumoperitoneum and Trendelenburg position.
   * Peak airway pressure exceeding 35 cm H2O
3. Patients with a history of allergy to lidocaine.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients scheduled for laparoscopic hysterectomy surgery.
Enrollment: 66 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Optic Nerve Sheath Diameter (ONSD) | 5 min before induction of anesthesia till 5 min after the closure of pneumoperitoneum
  ONSD at 5 min before induction of anesthesia in supine position (T1), 5 min after CO2 pneumoperitoneum in Trendelenburg position (T2), 30 min after CO2 pneumoperitoneum in Trendelenburg position (T3), 60 min after CO2 pneumoperitoneum in Trendelenburg position (T4) and 5 min after the closure of pneumoperitoneum in supine position (T5).

SECONDARY OUTCOMES:
Heart rate | 5 min before induction of anesthesia till 5 min after the closure of pneumoperitoneum
  Heart rate at 5 min before induction of anesthesia in supine position (T1), 5 min after CO2 pneumoperitoneum in Trendelenburg position (T2), 30 min after CO2 pneumoperitoneum in Trendelenburg position (T3), 60 min after CO2 pneumoperitoneum in Trendelenburg position (T4) and 5 min after the closure of pneumoperitoneum in supine position (T5).
Mean arterial blood pressure | 5 min before induction of anesthesia till 5 min after the closure of pneumoperitoneum
  Mean arterial blood pressure at 5 min before induction of anesthesia in supine position (T1), 5 min after CO2 pneumoperitoneum in Trendelenburg position (T2), 30 min after CO2 pneumoperitoneum in Trendelenburg position (T3), 60 min after CO2 pneumoperitoneum in Trendelenburg position (T4) and 5 min after the closure of pneumoperitoneum in supine position (T5).
The incidence of postoperative adverse reactions | Within 3 hours after surgery
  The incidence of adverse reactions, such as dizziness, postoperative nausea and vomiting (PONV) and postoperative headache (POHA) within 3 hours after surgery will be recorded in both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, ElGharbiaa, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP
Time Frame: After completion of the study
Access Criteria: The data will be available upon reasonable request from the corresponding author